CLINICAL TRIAL: NCT05236569
Title: Effectiveness and Safety of Intradermal Tranexamic Acid Injection as An Adjunctive Treatment for Melasma in Skin Type IV - V: A Double-Blind Randomized Controlled Trial
Brief Title: Effectiveness and Safety of Intradermal Tranexamic Acid Injection as An Adjunctive Treatment for Melasma in Skin Type IV - V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Vashty Amanda Hosfiar, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-11-1376
Record Dates: First submitted 2022-01-28; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Melasma
Keywords: melasma; tranexamic acid; modified melasma area and severity index; melanin index; erythema index
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomized to receive either 10 mg of intradermal tranexamic acid injection or placebo on one side of the face with 1:1 ratio. The allocation sequence was generated with a computer by an analyst.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation sequence was generated with a computer by an analyst. The allocation sequence was concealed from the investigators, care provider, outcomes assessor, and subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (Experimental): The intervention was 1 ml of 10 mg/ml of tranexamic acid solution which was given intradermally.
  Interventions: Drug: Tranexamic acid injection
- Placebo (Placebo Comparator): The placebo was 1 ml of 0.9% normal saline which was given intradermally.
  Interventions: Drug: Injection Water

INTERVENTIONS:
Drug: Tranexamic acid injection — The tranexamic acid injection was given intradermally to the facial skin
  Arms: Tranexamic acid
Drug: Injection Water — The 0.9% normal saline injection was given intradermally to the facial skin
  Arms: Placebo

SUMMARY:
A double-blind, randomized, split-face controlled trial of 34 female patients with melasma was conducted. All subject were randomized to receive either intradermal tranexamic acid or placebo injection on the right or the left side of their face.

DETAILED DESCRIPTION:
All subject were randomized to receive either 10 mg of intradermal tranexamic acid or placebo injection on the right or the left side of their face.

The primary outcome was improvement of melasma lesions assessed by modified Melasma Area and Severity Index (mMASI) score and mexameter examination which includes Melanin Index (MI) and Erythema Index (EI).

Measurements were done at baseline and every two weeks for twelve weeks. Additionally, side effects of therapy and subjects' satisfactory assessment with patient global assessment (PtGA) were also documented.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 60 years old
* Fitzpatrick skin type IV - V
* diagnosed with melasma

Exclusion Criteria:

* pregnancy and breastfeeding
* use of oral contraceptives within six months
* use of topical or systemic melasma therapy within two weeks
* history of superficial peeling within four weeks
* history of dermabrasion within six months
* use of photosensitizer drugs
* history of thrombosis or currently using antithrombotic or anticoagulant drugs
* history of TA allergy
* experiencing any COVID-19 symptoms

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Modified Melasma Area and Severity Index (mMASI) score | 12 weeks
  Reduction of mMASI score
Erythema Index | 12 weeks
  Reduction of erythema index
Melanin Index | 12 weeks
  Reduction of melanin index

SECONDARY OUTCOMES:
Side effects | 12 weeks
  Incidence of side effects
Subject's satisfaction | 12 weeks
  Satisfaction towards the treatment's results measured by patient global assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology and Venereology Clinic, Dr. Cipto Mangunkusumo National Central General Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No